CLINICAL TRIAL: NCT01984905
Title: Exploratory Study of Prognostic Factors in Aortic Dissection Type B: Role of Imaging (18F-FDG PET-Scan and Angioscan) and Biomarkers
Brief Title: Study of Prognostic Factors in Aortic Dissection Type B
Acronym: TEDAC
Status: Terminated | Type: Observational
Why Stopped: insufficient patient recruitment
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00209-36
Record Dates: First submitted 2013-10-25; First posted 2013-11-15 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Type B Aortic Dissection
Keywords: 18 FDG PET-scan; angioscan; aortic dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical outcomes of chronic type B aortic dissections are unknown, especially in case of false lumen expansion and risk of rupture. Data of literature give us some indications about prognosis. The 1-year survival rate is about 80%, but we deplore the 25% rate of mortality at 3 years despite follow-up.The only known predictive factors are the initial diameter of more than 4 cm and the persistence of a false lumen patent.However, actual means of follow-up do not allow to predict severe complications. The aim of the sudy is to propose a diagnostic and preventive strategy for the follow-up of chronic type B aortic dissections treated medically.

The primary objective is then to evaluate the prognostic role of 18-FDG-PET Scan in such patients in order to predict the risk of aortic diameter growth of more than 5 mm in 1 year and/or of an aortic dissections extension at 1 year. The secondary objectives are to evaluate the link between fibrosis biomarkers MMP et TIMP) and the results of imaging results (evolution of diameter and extension and results of PET-Scan imaging) Methods: 100 patients to be included in 3 years History of chronic type B aortic dissection, treated medically, evolving since more than 1 month and less than 5 years.

Expected results: Prognostic contribution of 18FDG-PET-Scan and biomarkers for the identification of patients at high risk of evolution. Elaboration of a decisional algorithm about follow-up modalities of chronic aortic dissections. Demonstration of a correlation between aortic diameter growth or aortic dissection extension and intensity of marker fixation with 18-FDG-PET-Scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Chronic type B aortic dissection, without surgical treatment
* Medically treated patient
* Medical treatment since more than 1 month and less than 5 years
* Aortic dissection localization : below left subclavian artery and alow femoral artery
* Affiliation to a social security system
* Patient who have given informed consent

Exclusion Criteria:

* History of malignant pathology
* Aortic dissection since less than 1 month or more than 5 years
* Inflammatory or infectious disease of the aorta
* Uncontrolled infectious disease
* Iodine Allergy
* Severe renal insufficiency (cockcroft clearance <30 mL/min)
* Patient under guardianship or curators
* Any associated medical or psychological condition wich could compromise the patient's ability to participate in the study
* Inability to be submitted to the study follow-up for geographical, social or psychological reasons
* Current pregnancy or lack of effective contraception during their reproductive years
* Suckle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from chronic type B aortic dissection (since more than 1 month and less than 5 years)and medically treated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10-25 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Correlation between the increase in the aortic diameter and the intensity of 18-FDG binding (Standard Uptake Value) at 1 year | 1 year

SECONDARY OUTCOMES:
Correlation between biomarkers of fibrosis and results of morphological and functional imaging | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ludovic BERGER, MD,PhD, Principal Investigator — Caen UH
Locations (1):
- Caen University Hospital, Caen, France